CLINICAL TRIAL: NCT06962761
Title: Impact of Vit D and Probiotic As a Supplementary Therapy in The Treatment of PatientWith Bronchial Asthma
Brief Title: the Effect of Use of Vit d and Probiotic as a Supplementaition in the Treatment of Bronchial Asthma in Patient Aged 6 to 50 Year and Its Effect in Decrasing Excerbation.
Acronym: asthma
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, abdelrahman ahmed mohamed ibrahim, resident doctor of chest department Al-Azhar university asyut, Al-Azhar University
Other Study IDs: MSC\AZ.AST\C11T019\29\227
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Probiotics

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- adult and children with bronchial asthma: 4 groups 2adult groups 1take the vitd and probiotic andregulartreatment of asthma and another take regulartreatment of asthma only 2 children groups 1take the vitd and probiotic andregulartreatment of asthma and another take regulartreatment of asthma only
  Interventions: Drug: Vit D

INTERVENTIONS:
Drug: Vit D — in this study we use a combination of vit d and probiotics
  Other Names: probiotics

SUMMARY:
the study of the effect of vit d and probiotic as suprplementaion in the treatment of patient with bonchial asthma and its effect in decreasing number of excerbation

DETAILED DESCRIPTION:
the study of the effect of vit d and probiotic as suprplementaion in the treatment of patient with bonchial asthma and its effect in decreasing number of excerbation

ELIGIBILITY:
Inclusion Criteria: patient wih bronchial asthma aged 6 to50years -

Exclusion Criteria: other comorbities

-

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: patient wih bronchial asthma
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
asthma control test | 3,6 and 12 months
  The ACT has five questions and assesses the frequency of shortness of breath and general asthma symptoms, the use of rescue medications, the effect of asthma on daily functioning, and an overall self-assessment of asthma control in the last four weeks. Scores range from 5 (poor control of asthma) to 25 (complete control of asthma), and high scores reflect greater degrees of asthma control. Asthma is classified as controlled if the score is greater than 19

CONTACTS AND LOCATIONS:
Locations (1):
- ALAzhar university hospital assiut, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol